CLINICAL TRIAL: NCT02583867
Title: Predictors of Depression Treatment Response to Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 052015-018
Record Dates: First submitted 2015-10-13; First posted 2015-10-22 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): Participants will complete an exercise dose of 15 kilocalories per kilogram of bodyweight per week (KKW). This is equivalent to approximately 150 minutes/week of aerobic exercise. This dose will be completed in at least 3 sessions per week for 12 weeks.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Subjects will engage in supervised exercise sessions for 12 weeks. Each week will consist of at least three exercise sessions with a total duration of weekly exercise of approximately 150 minutes.

SUMMARY:
50 subjects with Major Depressive Disorder who are not currently receiving treatment will be enrolled in a 12-week exercise program, supervised by a trained exercise interventionist.

DETAILED DESCRIPTION:
50 subjects with Major Depressive Disorder who are not currently receiving treatment will be enrolled in a 12-week exercise program, supervised by a trained exercise interventionist. Blood samples will be collected at baseline for analysis of inflammatory cytokines, as well as other potential biological predictors of treatment outcomes (i.e., BDNF). Assessments will gather data on potential clinical predictors of treatment outcomes (anxiety, stress, sleep). Assessments and sample collection will also occur at 3 time points during the treatment period (Weeks 4, 8, and 12) to identify mediators and correlates of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with MDD
2. Ages 18-65 will be included.
3. Ability to understand and willingness to provide written informed consent.
4. Willing to provide contact information.
5. Medical clearance with protocol-defined stress testing (in accordance with American College of Sports Medicine (ACSM) guidelines) from protocol approved medical personnel. Details of guidelines and related testing protocol are provided in the study Manual of Procedures.
6. Able to comprehend and communicate in English.

Exclusion Criteria:

1. Have a medical condition contraindicating exercise participation
2. Are currently physically active - defined as moderate intensity physical activity on 3 or more days per week for the last month
3. Currently receiving antidepressant medication treatment
4. Currently considered a high suicide risk and/or high risk for being unable to complete the study due to the need for psychiatric hospitalization, suicide attempts or suicidality, significant self-mutilation, or other self-injurious or destructive behavior based on the judgment of the site PI, medical personnel, or designee.
5. Pregnancy.
6. Current psychotic disorder. Other comorbid psychiatric diagnosis that, in the investigator's judgment, will pose a safety issue or make it difficult for the participant to understand or complete the intervention.
7. Anticipated circumstances over the 6-month course of the trial that would render the participant unlikely to complete the study in the judgment of the PI or designee.
8. Any reason not listed herein yet, determined by the PI, medical personnel, or designee that constitutes good clinical practice and that would in the opinion of the PI, medical personnel, or designee make participation in the study hazardous.
9. Are currently enrolled in another research study, and participation in that study contraindicates participation in the current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-12; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms | 12 weeks
  Depressive symptoms will be assessed using the clinician-rated Inventory for Depressive Symptomatology (IDS-C)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Rethorst, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States